CLINICAL TRIAL: NCT00274560
Title: A Multiple Dose Comparison of Tiotropium Inhalation Capsules and Salmeterol Inhalation Aerosol in a 12 Week, Randomized, Double-Blind, Double-Dummy Parallel Group Study in Patients With Chronic Obstructive Pulmonary Disease (COPD).
Brief Title: A Multiple Dose Comparison of Tiotropium Inhalation Capsules and Salmeterol Inhalation Aerosol.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 205.264
Record Dates: First submitted 2006-01-09; First posted 2006-01-11 (Estimated); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Tiotropium Bromide; Salmeterol Xinafoate

INTERVENTIONS:
Drug: Tiotropium
Drug: Salmeterol

SUMMARY:
The objective of the study was to evaluate the degree of improvement in lung function in patients with chronic obstructive pulmonary disease (COPD) after treatment with tiotropium inhalation capsules compared to salmeterol inhalation aerosol .

ELIGIBILITY:
Inclusion criteria:

* Ability to sign a written Informed Consent Form consistent with International Conference of Harmonization-Good Clinical Practice (ICH-GCP) guidelines prior to participation in the trial (i.e., prior to any study procedures, including any pre-study washout of medications).
* Age of 40 years or older.
* Smoking history of ≥10 pack-years.
* A diagnosis of relatively stable chronic obstructive pulmonary disease with an Forced expiratory volume in one second (FEV1) ≤60% of predicted normal and FEV1 ≤70% of Forced vital capacity (FVC).
* Ability to perform technically acceptable pulmonary function tests, and ability to maintain records during the study period as required in the protocol.
* Ability to inhale medication from the HandiHaler® and from a metered dose inhaler.

Exclusion criteria:

* Clinically significant diseases other than Chronic obstructive pulmonary disease (COPD). A clinically significant disease was defined as a disease or condition which, in the opinion of the investigator, could have put the patient at risk because of participation in the study or may have influenced either the results of the study or the patient's ability to participate in the study.
* Known moderate or severe renal insufficiency.
* A recent history (i.e., six months or less) of myocardial infarction.
* Unstable or life-threatening cardiac arrhythmias, including newly diagnosed, clinically relevant arrhythmia on the electrocardiogram (ECG) performed on Visit 1. Unstable arrhythmias included arrhythmias that required an intervention (i.e., hospitalization, cardioversion, pacemaker placement, and automatic implantable cardiac defibrillator (AICD) placement) or a change in drug therapy during the year preceding study enrollment.
* Hospitalization for heart failure during the past three years.
* History of life-threatening pulmonary obstruction, or a history of cystic fibrosis or clinically evident bronchiectasis.
* Other exclusion criteria apply.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 653 (Actual)
Dates: Start 2002-05-01 (Actual); Primary Completion 2003-03-27 (Actual)

PRIMARY OUTCOMES:
FEV1 area under the curve for the time period of 0 to 12 hours (FEV1 AUC0-12) | 12 weeks
peak FEV1 | 12 weeks

SECONDARY OUTCOMES:
Trough FEV1: Trough FEV1 was the FEV1 measured prior to dosing | 12 weeks
Trough and peak FVC and FVC AUC0-12 measured at the same times as FEV1 on each test day | 12 weeks
Individual FEV1 and FVC measurements at each timepoint | 12 weeks
Number (%) of patients with at least one exacerbation of COPD | 12 weeks
time to first exacerbation | 12 weeks
number of exacerbations | 12 weeks
number of exacerbation days | 12 weeks
Average daily occasions of rescue medication [albuterol (salbutamol)] use each week | 12 weeks
All adverse events | 12 weeks
Pulse rate measured in conjunction with spirometry | 12 weeks
Blood pressure (seated) measured in conjunction with spirometry | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim Study Coordinator, Study Chair — Boehringer Ingelheim
Locations (50):
- United States (20):
  - UAB Medical Center, Birmingham, Alabama
  - Boehringer Ingelheim Investigational Site, Jasper, Alabama
  - Boehringer Ingelheim Investigational Site, Phoenix, Arizona
  - Southern Arizona VA Health Care System, Tucson, Arizona
  - Boehringer Ingelheim Investigational Site, Fullerton, California
  - VA Greater Los angeles Health Care Systems, Sepulveda, California
  - Olive View UCLA Medical Center, Sylmar, California
  - Boehringer Ingelheim Investigational Site, Boulder, Colorado
  - Colorado Pulmonary Associates, Denver, Colorado
  - Boehringer Ingelheim Investigational Site, Wheat Ridge, Colorado
  - Boehringer Ingelheim Investigational Site, Melbourne, Florida
  - Boehringer Ingelheim Investigational Site, Pembroke Pines, Florida
  - University Medical Associates, LLP, Augusta, Georgia
  - Boehringer Ingelheim Investigational Site, Coeur d'Alene, Idaho
  - LSU MC-Sheveport, Shreveport, Louisiana
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - The Oregon Clinic, Portland, Oregon
  - Temple University School of Medicine, Philadelphia, Pennsylvania
  - Attention: Thomas D. Kaelin, Jr., D.O., Charleston, South Carolina
  - Boehringer Ingelheim Investigational Site, Houston, Texas
- Finland (3):
  - HEMO Oy Health Center, Lahti
  - Boehringer Ingelheim Investigational Site, Mikkeli
  - Boehringer Ingelheim Investigational Site, Oulu
- Greece (6):
  - Gen. Hosp. "Evangelismos",, Athens
  - Gen. Hosp. of Chest Diseases "Sotiria", Athens
  - Gen. Hosp. of Chest Diseases"Sotiria", Athens
  - University Hospital of Ioannina, Ioannina
  - General Hospital "Sismanoglio", 3rd Pneumonology Dpt, Maroussi, Athens
  - General Hospital "Papanicolaou",, Thessaloniki
- Italy (2):
  - Azienda Ospedaliera S. Martino, Genova
  - A.O. Pisana, Pisa
- Portugal (4):
  - Hospital de Santa Maria, Lisbon
  - Hospital Pulido Valente, Lisbon
  - Hospital de São João, Porto
  - Centro Hospitalar de Vila Nova de Gaia, Vila Nova de Gaia
- Sweden (7):
  - Lindesbergs lasarett, Lindesberg
  - Boehringer Ingelheim Investigational Site, Linköping
  - Vårdcentralen Brinken, Motala
  - Boehringer Ingelheim Investigational Site, Örebro
  - Boehringer Ingelheim Investigational Site, Stockholm
  - Fysiologlaboratoriet, Stockholm
  - Boehringer Ingelheim Investigational Site, Uppsala
- Turkey (Türkiye) (4):
  - Gazi Universitesi Tip Fakultesi, Ankara
  - Istanbul Universitesi Cerrahpasa Tip Fakültesi, Istanbul
  - Yedikule Gögüs Hastaliklari Hastanesi, Istanbul
  - Ege Universitesi Tip Fakultesi, Izmir
- United Kingdom (4):
  - Frenchay Healthcare NHS Trust, Bristol
  - Boehringer Ingelheim Investigational Site, Glasgow
  - West Middlesex University Hospital, Isleworth
  - Medicines Evaluation Unit, Manchester